CLINICAL TRIAL: NCT01771055
Title: Direct Peritoneal Resuscitation Effects in the Damage Control Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Jason Smith, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09.0178
Record Dates: First submitted 2013-01-11; First posted 2013-01-18 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Traumatic Injury
Keywords: Trauma; Hypovolemia
MeSH Terms: conditions — Wounds and Injuries; Hypovolemia | interventions — Galactose

STUDY DESIGN:
Intervention Model Description: Galactose versus standard care
Oversight: Data Monitoring Committee: No

ARMS (2):
- Galactose (Experimental): Galactose
  Interventions: Procedure: Galactose
- Standard resuscitation (Placebo Comparator): Standard surgical methods of controlling bleeding
  Interventions: Procedure: Standard surgical methods

INTERVENTIONS:
Procedure: Galactose — Galactose dripped into the abdomen after surgery
  Arms: Galactose
Procedure: Standard surgical methods
  Arms: Standard resuscitation

SUMMARY:
The purpose of this study is to find if direct peritoneal resuscitation helps blood flow through important organs in a person's body after they have had a traumatic injury with massive blood loss. Sometimes after severe injuries requiring operation, surgeons cannot close the muscles and skin of a patient's belly, because of swelling. This study will also try to find if direct peritoneal resuscitation decreases tissue swelling and allows for quicker closure of of a patient's belly.

DETAILED DESCRIPTION:
Standard methods of controlling bleeding and increasing blood flow to vital organs will be used. These methods include giving blood and fluids and surgically repairing the vessels that are causing the bleeding which are standard ways physicians treat injuries with massive blood loss. A drain (a small plastic tube) will be placed inside the belly.

Subjects will randomly (like flipping a coin) be placed into a group of patients who either get a sugar solution dripped into the belly after surgery or do not get this treatment. The drain will be used to drip a high glucose solution into the abdomen in patients be part of that group. The fluid will continue to be dripped into the belly until it is possible to close the skin and underlying layers.

ELIGIBILITY:
Inclusion Criteria:

* All trauma patients age 18 years or greater with massive blood loss
* Patients requiring a damage control procedure
* Traumatic injury within the last 24 hours

Exclusion Criteria:

* Patients who are pregnant
* Less than 18 years of age
* Known chronic renal disease
* Moribund

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Smith, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Standard of care without peritoneal resuscitation
- Direct Peritoneal Resuscitation: Subjects received standard operation plus direct peritoneal resuscitation after surgery
Period: Overall Study
Arm/Group | Control | Direct Peritoneal Resuscitation
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Resuscitation: Standard surgical methods of controlling bleeding
  Standard surgical methods
- Total: Total of all reporting groups
Arm/Group | Galactose | Standard Resuscitation | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 2 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Morbidity
Description: Evaluate the Number of participants with Morbidity receiving Direct Peritoneal Resuscitation versus those receiving standard care.
Time Frame: 1 Month
Measure: Number; unit: number of participants
Groups:
- Standard Resuscitation: Standard surgical methods of controlling bleeding
  Standard surgical methods without galactose
Arm/Group | Galactose | Standard Resuscitation
Number analyzed (Participants) | 3 | 4
number of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | Galactose | Standard Resuscitation
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No